CLINICAL TRIAL: NCT01848665
Title: The Influence of Cerebral Blood Flow and PETCO2 on Neuromuscular Function During Passive Heat Stress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Stephen Cheung, Professor, Brock University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: EEL 073.3
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Healthy Males; Neuromuscular Function
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Drug (Experimental): Indomethacin, 1.2 mg kg 1 dose
  Interventions: Drug: Indomethacin
- Placebo (Placebo Comparator): generic flour placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin
  Arms: Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
Increased core temperature (hyperthermia) has been associated with impaired neuromuscular performance; however, the mechanisms associated with these performance decrements and their potential synergies remain unclear. While the majority of research suggests that the observed fatigue is related to the central nervous system, the influence of changes in cerebral blood flow (CBF) and associated changes in cerebral alkalosis (estimated by end-tidal partial pressure of carbon dioxide; PETCO2) remains unexamined. In response to hyperthermia, humans hyperventilate as means of heat dissipation, resulting in a hypocapnia (reduced PETCO2) mediated decrease in CBF and consequently, cerebral alkalosis (increased cerebral pH). Previous research suggests that hyperventilation induces changes in neural excitability and synaptic transmission; however, it remains unclear if these changes are related to hypocapnia mediated decrease in CBF or decreased PETCO2 or both.

The purpose of the proposed research program is to examine the influence of changes in CBF and cerebral alkalosis on neuromuscular function during passive heat stress. The research project will consist of 3 separate experimental trials: (a) poikilocapnic hyperthermia (increased core temperature; decrease CBF; decrease PETCO2), (b) isocapnic hyperthermia (increased core temperature; no change CBF; no change PETCO2) and (c) isocapnic hyperthermia + indomethacin (increased core temperature; decrease CBF; no change PETCO2). During each manipulation, neuromuscular function will be evaluated and compared to baseline (normothermic) conditions using a repeated measures design.

It is hypothesized that changes in PETCO2 and therefore, changes in cerebral alkalosis will contribute to neuromuscular fatigue independent of changes in CBF or increases in core temperature.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 yrs old; healthy males

Exclusion Criteria:

* diagnosed medical condition; NSAID allergy; smoker; high altitude exposure; implants

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Resting motor threshold | Change from baseline 90-minutes
  Motor evoked potentials are recorded from muscles following transcranial magnetic stimulation of motor cortex. The resting motor threshold is defined as the minimum stimulation intensity required to elicit a motor evoked potential. Resting motor threshold will be quantified in millivolts.
H-Reflex Amplitude | Change from baseline 90-minutes
  The H-Reflex is an indirect measure of motor neuron excitability. Initially, a maximal M-wave (M-max) will be elicited by stimulating (1 ms in duration; 15 s between stimuli) the median nerve incrementally (2 V increments) until the largest waveform is observed. The peak-to-peak amplitude of this waveform is considered M-max. Using similar procedures as above, a sub-maximal M-wave of 5% M-max will be elicited and the amplitude of the resultant H-reflex (a small waveform observed following the submaximal M-wave) will be calculated. The amplitude of the H-reflex will be quantified in millivolts.
Maximal Voluntary Contraction | Change from baseline 90-minutes
  During maximal voluntary contraction (MVC) testing, the participants' right arm will be secured in a custom made device used to isolate forearm flexion and to measure force production by the flexor carpi radialis muscle. Participants will be asked to produce a 5-second MVC and will be verbally encouraged to maintain maximal force production throughout the duration of the contraction. MVC will be quantified as the maximum force production in newton meters.
H-Reflex latency | Change from baseline 90-minutes
  The H-Reflex is an indirect measure of motor neuron excitability. Initially, a maximal M-wave (M-max) will be elicited by stimulating (1 ms in duration; 15 s between stimuli) the median nerve incrementally (2 V increments) until the largest waveform is observed. The peak-to-peak amplitude of this waveform is considered M-max. Using similar procedures as above, a sub-maximal M-wave of 5% M-max will be elicited and the amplitude of the resultant H-reflex (a small waveform observed following the submaximal M-wave) will be calculated. The onset latency of the H-reflex will be quantified in milliseconds.
Voluntary Activation | change from baseline 90-minutes
  The level of neural drive to muscle during contraction is termed voluntary activation and will be estimated by interpolation of a single supramaximal motor evoked potential during the 5-second MVC contraction. If extra force is evoked by the 'superimposed' stimulus then either the stimulated axons were not all recruited voluntarily or they were discharging at sub-tetanic rates. Therefore, voluntary activation will be quantified as the amplitude of maximal voluntary force production, relative to the amplitude of the supramaximal MEP.

SECONDARY OUTCOMES:
Middle Cerebral Artery Blood Flow Velocity | Change from baseline 90-minutes
  Middle cerebral artery (MCA) blood flow velocity will be measured non-invasively by a 2-MHz transcranial Doppler (TCD) ultrasound probe, attached bilaterally to a comfortable headband and secured anterior to the zygomatic arch, rostral of the pinna. Doppler probes will be paced over the temporal windows (near the ear) and will remain in place throughout the duration of the experimental protocol. MCA velocity will be quantified in cm/s.
Blood Pressure | Change from baseline 90-minutes
  Beat by beat blood pressure will be calculated from the blood pressure waveform using finger photoplethysmography (Nexfin, bmeye), with a finger cuff placed directly over the middle finger on the left hand. Blood pressure will be quantified in mmHg.
Heart rate | Change from baseline 90-minutes
  Heart rate will be measured by electrocardiogram. Heart rate will be quantified in beats per minute.
End-tidal Gas concentrations | change from baseline 90-minutes
  The end-tidal concentrations of oxygen and carbon dioxide will be measured and reported in mmHg.
Rectal Temperature | change from baseline 90-minutes
  Rectal temperature will be measured in degrees Celsius
Skin Temperature | change from baseline 90-minutes
  skin temperature will be measured in degrees Celsius

CONTACTS AND LOCATIONS:
Locations (1):
- Brock University, St. Catharines, Ontario, Canada